CLINICAL TRIAL: NCT06343116
Title: Randomized Double-blind, Placebo-controlled, Multicenter Clinical Study of Nimotuzumab Combined With Trifluridine/Tipiracil in Third-line and Beyond for the Treatment of Metastatic Colorectal Cancer
Brief Title: Nimotuzumab Combined With Trifluridine/Tipiracil in the Treatment of Refractory Metastatic Colorectal Cancer
Acronym: NOTABLE-308
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BPL-Nim-CRC-3001
Record Dates: First submitted 2024-03-18; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Refractory Metastatic Colorectal Cancer
Keywords: Nimotuzumab; trifluridine/tipiracil; metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — nimotuzumab; trifluridine tipiracil drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Nimotuzumab will be administered weekly (dose of nimotuzumab depends on part A). Trifluridine/tipiracil will be administered (35 mg/m2) twice daily, 5 days a week, with 2 days of rest, for 2 weeks, followed by a 14-day rest. Treatment will continue until disease progression, unacceptable toxicity, withdrawal of consent or death due to any cause.
  Interventions: Drug: Nimotuzumab injection; Drug: Trifluridine/tipiracil
- control group (Placebo Comparator): Placebo will be administered weekly (dose of placebo depends on part A). Trifluridine/tipiracil will be administered (35 mg/m2) twice daily, 5 days a week, with 2 days of rest, for 2 weeks, followed by a 14-day rest. Treatment will continue until disease progression, unacceptable toxicity, withdrawal of consent or death due to any cause.
  Interventions: Drug: Placebo; Drug: Trifluridine/tipiracil

INTERVENTIONS:
Drug: Nimotuzumab injection — Nimotuzumab will be administered weekly (dose of nimotuzumab depends on part A) until disease progression, unacceptable toxicity, withdrawal of consent or death due to any cause.
  Other Names: Taixinsheng
  Arms: experimental group
Drug: Placebo — Placebo will be administered weekly (dose of placebo depends on part A) until disease progression, unacceptable toxicity, withdrawal of consent or death due to any cause.
  Arms: control group
Drug: Trifluridine/tipiracil — Trifluridine/tipiracil will be administered (35 mg/m2) twice daily, 5 days a week, with 2 days of rest, for 2 weeks, followed by a 14-day rest.

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter study. The main purpose of the study is to evaluate the clinical efficacy and safety of nimotuzumab combined with trifluridine/tipiracil in third-line and beyond for the treatment of metastatic colorectal cancer (mCRC). This study planned to be divided into two parts: Part A and Part B. Part A (safety run-in) with a 3 + 3 study design, which primary endpoint is safety; Part B (main study) with a prospective, randomized, double-blind, placebo-controlled design, which primary endpoint is overall survival (OS).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter study. The main purpose of the study is to evaluate the clinical efficacy and safety of nimotuzumab combined with trifluridine/tipiracil in third-line and beyond for the treatment of metastatic colorectal cancer (mCRC). This study planned to be divided into two parts: Part A and Part B. Part A is a dose escalation study, and two dose levels are set up in terms of the dose of nimotuzumab (dose level 1: nimotuzumab 400 mg weekly; dose level 2: nimotuzumab 600 mg weekly), while the dose of trifluridine/tipiracil remains unchanged. The aim of this part is to investigate the safety of combination therapy and ensure the dose of nimotuzumab in Part B. After completed the safety-run-in of Part A, Part B can be started. In Part B (main study), a prospective, randomized, double-blind, placebo-controlled design is proposed. Patients of this part will be stratified by tumor site (left half of colorectal vs right half of colon), age (less than 65 years old vs 65 years old or older) and number of metastases (<3 vs ≥3) and randomly divided into experimental group (nimotuzumab plus trifluridine/tipiracil) and control group (placebo plus trifluridine/tipiracil) at a ratio of 2:1. Treatment will continue until disease progression or intolerable toxicity or withdrawal of consent. In part B, the primary endpoint is overall survival (OS); the secondary endpoint included: Progression free survival (PFS), time to progress (TTP), overall response rate (ORR), disease control rate (DCR), duration of response (DoR), quality of life (QoL), etc.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, gender unlimited;
2. Histologically or cytologically confirmed diagnosis of colorectal cancer (CRC);
3. Metastatic colorectal cancer, disease progression after previous second-line or above standard therapy;
4. Efficacy of previous line therapy containing an anti-EGFR agent (panitumumab or cetuximab) with complete or partial response, or disease stable; and more than 4 months from last dose of anti-EGFR agent administered before randomization;
5. MSS/pMMR status detected by IHC or PCR;
6. RAS and BRAF wild-type status;
7. ECOG Performance Status 0-1;
8. Measurable disease according to RECIST criteria v1.1;
9. Life expectancy of at least 3 months;
10. Adequate organ and bone marrow function, defined as follows: hemoglobin≥9.0 g/dL; absolute neutrophil count (ANC)≥1.5×10^9/L; white Blood Cell Count≥4×10^9/L;platelets≥100×10^9/L; serum total bilirubin (TBIL)≤1.5×ULN; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of normal (ULN), patients with liver metastases should be ≤ 5 times the ULN; serum creatinine≤1.5×ULN or estimated creatinine clearance > 60 mL/min;
11. Women of childbearing age should have a negative result of serum HCG or urine pregnancy tests within 72 hours prior to randomization (Postmenopausal women who have had amenorrhea for at least 12 months are considered sterile and women known to have had tubal ligation are not required to undergo pregnancy tests) ;
12. Good compliance and signed informed consent.

Exclusion Criteria:

1. Had other malignancies within the past 5 years or at the same time (exceptions include: cured thyroid cancer, non-melanoma skin cancer, carcinoma in situ of the cervix, stage I ductal carcinoma in situ, stage I endometrial cancer or other solid tumors, and effectively treated lymphoma with no evidence of disease for more than 5 years);
2. Has a serious underlying medical condition that makes it impossible to safely administer the trial treatment. Including but not limited to active infections requiring systemic medication: compensatory heart failure (NYHA grade III and IV), unstable angina, and acute myocardial infarction within 3 months prior to enrollment;
3. Patients who received trifluridine/tipiracil or treated with EGFR monoclonal antibody or EGFR tyrosine kinase inhibitor within four months;
4. Known allergy to prescription or any component of the prescription used in this study;
5. Women who are pregnant or are breastfeeding;
6. Has brain metastases or any symptoms of brain metastases
7. Factors that significantly affect oral drug absorption, such as dysphagia, chronic diarrhea, gastrointestinal obstruction, etc; Uncontrolled Crohn's disease or ulcerative colitis;
8. Participated in other clinical trials within 4 weeks;
9. With HIV, HPV, or syphilis infection, or active hepatitis (hepatitis B, hepatitis C)
10. Other reasons that are not suitable to participate in this study according to the researcher's judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) | Up to 18 months
  The primary endpoint is overall survival (OS, defined as from randomization to death due to any cause).
dose-limiting toxicity (DLT) | Up to 4 weeks for each participant in part A
  DLTs at the end of the 4 weeks' treatment in part A (safety run-in).

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to 18 months
  PFS, defined as from randomization to disease progression or all-cause death. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
time to progress (TTP) | Up to 18 months
  TTP, defined as from randomization to the first observation of disease progression. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
overall response rate (ORR) | Up to 18 months
  Objective response rate (ORR), including complete response (CR) and partial response (PR). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT/MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), at least a 30% decrease in the sum of the longest diameter of target lesions.
disease control rate (DCR) | Up to 18 months
  Disease control rate (DCR), including complete response (CR) and partial response (PR) and stable disease(SD). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT/MRI: CR, disappearance of all target lesions; PR, at least a 30% decrease in the sum of the longest diameter of target lesions.
  SD, neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD (PD, defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions).
duration of response (DoR) | Up to 18 months
  Duration of response (DoR) is defined as the period from the first evaluation of complete response (CR) and partial response (PR) to the first evaluation of disease progression or all-cause death.
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC-QLQ-C30) | Up to 18 months
  Quality of Life will be evaluated by European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC-QLQ-C30). The scale assesses symptoms, functionality, and overall health status/life quality. Each item is transformed to a 0-100 scale according to a standardized scoring procedure. Higher scores indicate more severe symptoms, while in the functionality and overall health status/life quality sections, higher scores signify better conditions.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Colorectal Cancer 29 (EORTC-QLQ-CR29) | Up to 18 months
  Quality of Life will also be evaluated by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Colorectal Cancer 29 (EORTC-QLQ-CR29). EORTC-QLQ-CR29 is a supplementary questionnaire module to be employed in conjunction with the Quality of Life Questionnaire Core 30 (QLQ-C30). All of the scales and single-item measures range in score from 0 to 100. A high score for the functional scale and functional single-items represents a high level of functioning, whereas a high score for the symptom scales and symptom single-items represents a high level of symptomatology or problems.
Adverse Events | Up to 18 months
  Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.

OTHER OUTCOMES:
tumor-related markers | Up to 18 months
  To explore the influence of tumor-related markers (such as EGFR, p53, etc.) on prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Study Chair — Peking University Cancer Hospital & Institute